CLINICAL TRIAL: NCT04040439
Title: Precedex(Registered) Intravenous Solution Special Investigation (in Pediatric Patients)
Brief Title: Precedex Special Investigation (in Pediatric Patients)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Maruishi Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: C0801023
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Results first posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-06

CONDITIONS: Sedation
Keywords: Precedex;; Dexmedetomidine Hydrochloride;; Sedation;; intensive care;; pediatric
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dexmedetomidine Hydrochloride: Pediatric patients (45 weeks corrected gestational age to <18 years old) administered Precedex (Dexmedetomidine Hydrochloride) for "sedation during and after mechanical ventilation in the intensive care setting"
  Interventions: Drug: Dexmedetomidine Hydrochloride

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — [Sedation during and after mechanical ventilation in the intensive care setting] For pediatric patients ages of 6 years and over, dexmedetomidine is usually administrated by continuous intravenous (IV) infusion of at a rate of 0.2 μg/kg/hr, following by continuous infusion at a range of 0.2 to 1.0 μg/kg/hr adjusted to achieve the optimal level of sedation depending on the patient's condition.
  For pediatric patients with corrected gestational ages (gestational age + postnatal age) of 45 weeks to under 6 years, dexmedetomidine is usually administrated by continuous IV infusion at a rate of 0.2 μg/kg/hr, following by continuous infusion at a range of 0.2 to 1.4 μg/kg/hr adjusted to achieve the optimal level of sedation depending on the patient's condition. The dosing rate could be decreased according to the patient's condition as appropriate.
  Other Names: Precedex

SUMMARY:
Secondary Data Collection:To confirm the safety and effectiveness profiles under the actual medical practice of Precedex in Japan.

DETAILED DESCRIPTION:
To assess the data, including safety profile, of Precedex Intravenous Solution administered for "sedation during and after mechanical ventilation in the intensive care setting" in pediatric patients under actual medical practice in Japan.

Maruishi Pharmaceutical Co., Ltd. and Pfizer Japan Inc. will collect 50 subjects each.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (45 weeks corrected gestational age to <18 years old) administered this drug for "sedation during and after mechanical ventilation in the intensive care setting.

Exclusion Criteria:

* No exclusion criteria is set out in this study.

Ages: 45 Weeks to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients (45 weeks corrected gestational age to <18 years old) administered this drug for "sedation during and after mechanical ventilation in the intensive care setting"
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Japan Local Country Office, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0801023

RESULTS

PARTICIPANT FLOW:
Groups:
- PRECEDEX INTRAVENOUS SOLUTION (Dexmedetomidine Hydrochloride): Pediatric patients (45 weeks corrected gestational age to <18 years old) administered Precedex for sedation during and after mechanical ventilation in the intensive care setting as indicated in the approved local product document were observed from the start of administration (hour 0) to the discharge from the intensive care unit (ICU) (up to Month 33, at the longest). The dosage can be adjusted as per physician's discretion.
  *IC=Informed Consent
Period: Overall Study
Arm/Group | PRECEDEX INTRAVENOUS SOLUTION (Dexmedetomidine Hydrochloride)
Started | 111
Completed | 98
Not Completed | 13
Not completed — Invalid registration | 11
Not completed — No IC* on publication of study results | 2

BASELINE CHARACTERISTICS:
Population: A total of 111 participants were enrolled in this study. Of the 111 participants who were enrolled and completed the study, 13 participants were excluded from the safety analysis population due to invalid registration (11 participants) and no informed consent on publication of study results (2 participants). Overall, the safety analysis set comprised of 98 participants.
Groups:
- PRECEDEX INTRAVENOUS SOLUTION (Dexmedetomidine Hydrochloride): Pediatric patients (45 weeks corrected gestational age to <18 years old) administered Precedex for sedation during and after mechanical ventilation in the intensive care setting as indicated in the approved local product document were observed from the start of administration (hour 0) to the discharge from the intensive care unit (ICU) (up to Month 33, at the longest). The dosage can be adjusted as per physician's discretion.
Arm/Group | PRECEDEX INTRAVENOUS SOLUTION (Dexmedetomidine Hydrochloride)
Number analyzed (Participants) | 98
Age, Customized [Number; unit: Participants]
  ≥45 weeks of corrected gestational age to <12 months of age | 35
  ≥12 to <24 months of age | 14
  ≥2 to <6 years | 27
  ≥6 to <18 years | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to Precedex in a participant who received Precedex. A serious ADR was an ADR resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to Precedex was assessed by the physician.
Time Frame: From the start of administration of Precedex (hour 0) to the discharge from the intensive care unit (ICU) (up to Month 33, at the longest).
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and had received Precedex at least once. Participants with invalid registration or without informed consent were excluded.
Measure: Number; unit: Participants
Arm/Group | PRECEDEX INTRAVENOUS SOLUTION (Dexmedetomidine Hydrochloride)
Number analyzed (Participants) | 98
Participants
  ADR | 9
  Serious ADR | 2

2. Secondary Outcome: Percentage of Participants Who Were Evaluated as Effective (Responders) by the Physician
Description: Overall effectiveness of Precedex was evaluated at the end of Precedex administration by the physician. Clinical effectiveness was evaluated as effective, not effective, or indeterminate by the physician. Clinical effectiveness proportion was defined as the proportion of responders divided by the total number of responders and non-responders.
Time Frame: At the end of administration of Precedex (up to Month 33, at the longest)
Population: The effectiveness analysis set comprised of participants in the safety analysis set who had effectiveness evaluation by the physician at the end of Precedex administration. Participants who received Precedex for an out-of-scope indication, or those who received inadequate duration or dose of Precedex were excluded.
Measure: Number; unit: Percentage of participants
Arm/Group | PRECEDEX INTRAVENOUS SOLUTION (Dexmedetomidine Hydrochloride)
Number analyzed (Participants) | 76
Percentage of participants
  Effective | 100.0
  Not effective | 0.0
  Indeterminate | 0.0

ADVERSE EVENTS:
Time Frame: From the start of administration of Precedex (hour 0) to the discharge from the intensive care unit (ICU) (up to Month 33, at the longest).
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | PRECEDEX INTRAVENOUS SOLUTION (Dexmedetomidine Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 1/98
Serious Adverse Events (participants affected / at risk) | 4/98
Other Adverse Events (participants affected / at risk) | 8/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRECEDEX INTRAVENOUS SOLUTION (Dexmedetomidine Hydrochloride) (N=98)
Cardiac arrest (Cardiac disorders) | 2
Multiple organ dysfunction syndrome (Gastrointestinal disorders) | 1
Status epilepticus (Nervous system disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRECEDEX INTRAVENOUS SOLUTION (Dexmedetomidine Hydrochloride) (N=98)
Bradycardia (Cardiac disorders) | 2
Junctional ectopic tachycardia (Cardiac disorders) | 1
Pyrexia (General disorders) | 1
Blood pressure decreased (Investigations) | 2
Oxygen saturation decreased (Investigations) | 1
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/39/NCT04040439/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT04040439/SAP_001.pdf